CLINICAL TRIAL: NCT02326220
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Alirocumab in Patients With Heterozygous Familial Hypercholesterolemia Undergoing Lipid Apheresis Therapy
Brief Title: Study of Alirocumab (REGN727/SAR236553) in Patients With Heterozygous Familial Hypercholesterolemia (HeFH) Undergoing Low-density Lipoprotein (LDL) Apheresis Therapy
Acronym: ODYSSEY ESCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1216
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Heterozygous Familial Hypercholesterolemia
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Q2W (Double Blind Period) (Experimental): Placebo (for alirocumab) subcutaneous (SC) injection Q2W up to Week 16.
  Interventions: Drug: Placebo
- Alirocumab 150 mg Q2W (Double Blind Period) (Experimental): Alirocumab 150 mg SC injection Q2W up to Week 16.
  Interventions: Drug: Alirocumab
- Alirocumab 150 Q2W (Open Label Treatment Period) (Experimental): Alirocumab 150 mg SC injection Q2W starting from Week 18 up to Week 76.
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo Q2W (Double Blind Period)
Drug: Alirocumab
  Other Names: REGN727; SAR236553; Praluent®
  Arms: Alirocumab 150 Q2W (Open Label Treatment Period); Alirocumab 150 mg Q2W (Double Blind Period)

SUMMARY:
The primary objective of the study is to evaluate the effect of alirocumab 150 mg every 2 weeks (Q2W) in comparison with placebo on the frequency of low-density lipoprotein (LDL) apheresis treatments in participants with heterozygous familial hypercholesterolemia (HeFH) undergoing weekly or bi-weekly LDL apheresis therapy.

DETAILED DESCRIPTION:
LDL apheresis removes low-density lipoproteins (LDL) that transport cholesterol in the plasma portion of the blood. This treatment is mainly used for familial hypercholesterolemia, but can be used in other rare diseases. Familial hypercholesterolemia (HeFH) is an inherited genetic condition that causes accumulation of cholesterol in the blood, which can lead to atherosclerosis and heart disease. This treatment is recommended for patients who do not respond to dietary and/or medication control of LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age at the time of the screening visit
2. Diagnosis of HeFH (Heterozygous familial hypercholesterolemia)
3. Currently undergoing LDL (low-density lipoprotein) apheresis therapy QW (weekly) or Q2W (every 2 weeks) or at least 8 weeks prior to the screening visit

Exclusion Criteria:

1. Homozygous FH (familial hypercholesterolemia)
2. Background medical LMT (lipid-modifying therapy) (if applicable) that has not been stable for at least 8 weeks prior to the screening visit
3. LDL apheresis schedule/ apheresis settings that have not been stable for at least 8 weeks prior to the screening visit
4. An LDL apheresis schedule other than QW to Q2W
5. Initiation of a new exercise program or exercise that has not remained stable within 8 weeks prior to the screening visit (week -2)
6. Initiation of a new diet or a diet that has not been stable within 8 weeks prior to the screening visit (week -2)
7. Use of nutraceuticals or over-the-counter therapies known to affect lipids, at a dose/amount that has not been stable for at least 8 weeks prior to the screening visit (week -2), or between the screening and randomization visit
8. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins
9. Known history of a positive test for human immunodeficiency virus
10. Use of any active investigational drugs within 1 month or 5 half-lives of screening, whichever is longer
11. Patients who have been treated with at least 1 dose of alirocumab or any other anti-PCSK9 monoclonal antibody in any other clinical studies
12. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (13):
- United States (7):
  - Aurora, Colorado
  - Hartford, Connecticut
  - Kansas City, Kansas
  - Scarborough, Maine
  - Rochester, Minnesota
  - Portland, Oregon
  - Philadelphia, Pennsylvania
- Germany (6):
  - Dresden, Saxony
  - Berlin
  - Göttingen
  - Muenchen (2 Locations)
  - Passau
  - Rostock

REFERENCES:
- [Background] Moriarty PM, Parhofer KG, Babirak SP, Cornier MA, Duell PB, Hohenstein B, Leebmann J, Ramlow W, Schettler V, Simha V, Steinhagen-Thiessen E, Thompson PD, Vogt A, von Stritzky B, Du Y, Manvelian G. Alirocumab in patients with heterozygous familial hypercholesterolaemia undergoing lipoprotein apheresis: the ODYSSEY ESCAPE trial. Eur Heart J. 2016 Dec 21;37(48):3588-3595. doi: 10.1093/eurheartj/ehw388. Epub 2016 Aug 29. PMID 27572070
- [Derived] Moriarty PM, Parhofer KG, Babirak SP, deGoma E, Duell PB, Hohenstein B, Ramlow W, Simha V, Steinhagen-Thiessen E, Thompson PD, Vogt A, von Stritzky B, Du Y, Manvelian G. Alirocumab in patients with heterozygous familial hypercholesterolemia undergoing lipoprotein apheresis: Rationale and design of the ODYSSEY ESCAPE trial. J Clin Lipidol. 2016 May-Jun;10(3):627-34. doi: 10.1016/j.jacl.2016.02.003. Epub 2016 Feb 18. PMID 27206951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany and the United States between 09 Mar 2015 and 20 Apr 2016. A total of 76 participants were screened, of which 62 were enrolled and randomized in the study.
Pre-assignment Details: Randomization was stratified according to the frequency of the apheresis procedure (every 7 or 14 days) and lipoprotein (a) (Lp [a]) levels (normal or elevated). Assignment to treatment arms was done using an Interactive Voice/Web Response System in 1:2 ratio to placebo or alirocumab 150 mg Q2W.
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) subcutaneous (SC) injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment. (Participants undergoing LDL apheresis therapy every 1 or 2 weeks were enrolled in this study while maintaining background lipid modifying therapy (LMT) treatment throughout the study. All participants were being treated with the maximally tolerated clinically-relevant LMT).
- Alirocumab 150 mg Q2W (Double Blind Period): Alirocumab 150 mg SC injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment. (Participants undergoing LDL apheresis therapy every 1 or 2 weeks were enrolled in this study while maintaining background lipid modifying therapy (LMT) treatment throughout the study. All participants were being treated with the maximally tolerated clinically-relevant LMT).
- Alirocumab 150 Q2W (Open Label Treatment Period): Alirocumab 150 mg SC injection Q2W starting from Week 18 up to Week 76 or until alirocumab became commercially available in the subject's country, whichever occurred first. Apheresis treatment not required in the open-label treatment period and could be stopped or continued at the investigator's discretion. (All participants were being treated with the maximally tolerated clinically-relevant LMT.)
Period: Double-blind Treatment Period
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period) | Alirocumab 150 Q2W (Open Label Treatment Period)
Started | 21 (Out of 21 participants, 9 participants entered in open label treatment period) | 41 (Out of 41 participants, 20 participants entered in open label treatment period.) | 0
Completed | 20 | 37 | 0
Not Completed | 1 | 4 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Open-label Treatment Period
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period) | Alirocumab 150 Q2W (Open Label Treatment Period)
Started (Open-label available to participants in a country in which alirocumab was not commercially available) | 0 | 0 | 29 (29 participants: 9 from Placebo and 20 from Alirocumab 150 mg arm entered in open-label period.)
Completed | 0 | 0 | 27
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) SC injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment. (Participants undergoing LDL apheresis therapy every 1 or 2 weeks were enrolled in this study while maintaining background lipid modifying therapy (LMT) treatment throughout the study. All participants were being treated with the maximally tolerated clinically-relevant LMT).
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period) | Total
Number analyzed (Participants) | 21 | 41 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10.5) | 59.5 (9.2) | 58.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 10 | 26 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 41 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 21 | 39 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Frequency in which participants are undergoing LDL apheresis [Number; unit: Treatments] — LDL apheresis removes low-density lipoproteins (LDL) that transport cholesterol in the plasma portion of the blood. This treatment is mainly used for familial hypercholesterolemia, but can be used in other rare diseases. Familial hypercholesterolemia is an inherited genetic condition that causes accumulation of cholesterol in the blood, which can lead to atherosclerosis and heart disease. This treatment is recommended for patients who do not respond to dietary and/or medication control of LDL cholesterol.
  Treatments
    Every week | 9 | 18 | 27
    Every 2 weeks | 12 | 23 | 35
Calculated low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 191.6 (68.9) | 175.1 (54.6) | 180.7 (59.7)
Measured LDL-C [Mean (Standard Deviation); unit: mg/dL] | 195.0 (66.9) | 174.0 (51.4) | 181.1 (57.4)
Non-high-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 224.5 (68.0) | 210.3 (62.8) | 215.1 (64.4)
Total-cholesterol (Total-C) [Mean (Standard Deviation); unit: mg/dL] | 272.3 (73.6) | 256.9 (60.6) | 262.1 (65.1)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 47.8 (17.3) | 46.6 (16.2) | 47.0 (16.4)
Triglycerides (TGs) [Mean (Standard Deviation); unit: mg/dL] | 164.4 (61.4) | 176.0 (87.2) | 172.1 (79.0)
Lipoprotein a [Lp(a)] [Mean (Standard Deviation); unit: mg/dL] | 45.7 (49.5) | 43.0 (54.5) | 43.9 (52.4)
Apolipoprotein B (Apo-B) [Mean (Standard Deviation); unit: mg/dL] | 145.8 (34.0) | 135.2 (36.4) | 138.8 (35.7)
Apolipoprotein A1 (Apo-A1) [Mean (Standard Deviation); unit: mg/dL] | 145.8 (32.5) | 140.1 (25.5) | 142.1 (27.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Standardized Rate of Apheresis Treatments From Week 7 to Week 18
Description: Rate of apheresis treatments were normalized by the number of planned apheresis treatments according to each participant's established schedule at screening, week -10 to week -2. The normalized rate of apheresis was defined for each participant as the number of actual apheresis treatments received from week 7 to week 18 divided by the number of planned apheresis treatments per randomization strata at baseline (6 for Q2W and 12 for QW).
Time Frame: Week 7 to Week 18 (before start of open-label treatment)
Population: Primary intent-to-treat (ITT) population defined as all randomized participants and were analyzed according to the treatment group allocated by randomization.
Measure: Mean (Standard Deviation); unit: Treatments
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) subcutaneous (SC) injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment.
- Alirocumab 150 mg Q2W (Double Blind Period): Alirocumab 150 mg SC injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment.
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Treatments | 0.806 (0.191) | 0.128 (0.242)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); Analysis was performed using the ranked analysis of covariance (ANCOVA) model with baseline frequency of the apheresis procedure (QW or Q2W) and Lp(a) levels (normal or elevated) as fixed effect and the baseline LDL-C level as a covariate. Hodges-Lehmann estimator of median difference (median of all pairwise differences; CI is Moses distribution free CI. p-value is derived from the rank-based ANCOVA model. The model includes the baseline LDL-C value and stratification factors per IVRS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; H-L estimate of median difference = 0.750, 95% CI 2-sided [0.667 to 0.833] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C (Pre-apheresis) at Week 6
Description: Adjusted Least-squares (LS) means and standard errors at Week 6 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 2 to Week 18 regardless of status on or off-treatment were used in the model (ITT analysis).
Time Frame: Baseline and at Week 6
Population: Analysis was performed on ITT population that included all randomized particpants with baseline and at least one post-baseline pre-apheresis calculated LDL-C value up to week 6, analyzed according to the treatment group allocated by randomization.
Measure: Least Squares Mean (Standard Error); unit: percent change in mmol/L
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) SC injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or bi-weekly) until Week 6, then it was adjusted according to the response to treatment.
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percent change in mmol/L | 1.6 (3.1) | -53.7 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; MMRM: Mixed-effect model with repeated measures; Least Square (LS) Mean Difference = -55.3, 95% CI 2-sided [-63.0 to -47.5], Standard Error of Mean 3.9 — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

3. Secondary Outcome: Change in Standardized Rate of Apheresis Treatments From Week 15 to Week 18
Description: Rate of apheresis treatments were normalized by the rate by the number of actual apheresis treatments according to received from week 15 to week 18 divided by the planned apheresis treatments per randomization strata at baseline (2 for Q2W and 4 for QW). Only legitimate apheresis treatment skipping per point-of-care LDL-C value is counted as "apheresis not occurred". Missing apheresis treatment information (any reason) from week 7 to week 18 is assigned an outcome of the apheresis treatment occurred at the visit (i.e. impute 1 apheresis treatment for that visit).
Time Frame: Week 15 up to Week 18 (before the start of open-label treatment dose)
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: Treatments
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Treatments | 0.774 (0.315) | 0.165 (0.334)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < .0001, ANCOVA — Threshold for significance at 0.05 level; H-L estimate of median difference = 0.500, 95% CI 2-sided [0.500 to 1.000] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) (Pre-apheresis) to Week 6
Description: Adjusted LS means and standard errors at Week 6 were obtained from MMRM to account for missing data. All available post-baseline data from Week 2 (pre-apheresis) to Week 18 (pre-apheresis) regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 1.2 (3) | -42.8 (2.1)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -44, 95% CI 2-sided [-51.3 to -36.6] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

5. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) (Pre-apheresis) to Week 6
Description: as for outcome 4
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) SC injection Q2W up to Week 16. Apheresis frequency was fixed (weekly or biweekly) until Week 6, then it was adjusted according to the response to treatment.
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 2.8 (2.9) | -47.1 (2.1)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -50, 95% CI 2-sided [-57.3 to -42.7] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Pre-apheresis) to Week 6
Description: as for outcome 4
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 3.1 (2.5) | -36.4 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = -39.4, 95% CI 2-sided [-45.6 to -33.2] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A (Apo A1) (Pre-apheresis) to Week 6
Description: as for outcome 4
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 0 (3.3) | 4.2 (2.4)
Statistical Analysis 1: Comparison: Placebo Q2W (Double Blind Period) vs Alirocumab 150 mg Q2W (Double Blind Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3012, MMRM — Threshold for significance at 0.05 level; LS Mean Difference = 4.2, 95% CI 2-sided [-3.9 to 12.3] — Alirocumab 150 mg Q2W (Double Blind Period) vs. Placebo Q2W (Double Blind Period)

8. Secondary Outcome: Percentage of Participants With At Least (>=) 30% Reduction in Calculated LDL-C (Pre-apheresis) at Week 6
Description: Percentage of participants at Week 6 was obtained from a last observation carried forward (LOCF) model for handling of missing data. All available post-baseline data regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percentage of participants | 4.8 | 95.1

9. Secondary Outcome: Percentage of Participants With At Least (>=) 50% Reduction in Calculated LDL-C (Pre-apheresis) at Week 6
Description: Percentage of participants at Week 6 was obtained from LOCF model for handling of missing data. All available post-baseline data regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percentage of participants | 0 | 63.4

10. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C (Pre-Apheresis) to Week 18
Description: Adjusted LS means and standard errors at Week 18 were obtained from MMRM to account for missing data. All available post-baseline data from Week 2 (pre-apheresis) to Week 18 (pre-apheresis) regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 4 (6.2) | -42.3 (4.5)

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) (Pre-apheresis) to Week 18
Description: as for outcome 10
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percent change | 1.7 (4.8) | -33.8 (3.5)

12. Secondary Outcome: Percent Change From Baseline in Non-HDL-C (Pre-apheresis) to Week 18
Description: as for outcome 10
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 4.7 (5.6) | -35.7 (4.1)

13. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Pre-apheresis) to Week 18
Description: as for outcome 10
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 4.7 (4.7) | -27.1 (3.4)

14. Secondary Outcome: Percent Change From Baseline in Apo A1 (Pre-apheresis) to Week 18
Description: as for outcome 10
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | -0.7 (3.4) | 7.8 (2.4)

15. Secondary Outcome: Percentage of Participants With At Least (>=) 30% Reduction in Calculated LDL-C (Pre-apheresis) at Week 18
Description: Percentage of participants at Week 18 was obtained from LOCF model for handling of missing data. All available post-baseline data regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percentage of participants | 0 | 65.9

16. Secondary Outcome: Percentage of Participants With At Least (>=) 50% Reduction in Calculated LDL-C (Pre-apheresis) at Week 18
Description: as for outcome 15
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percentage of participants | 0 | 43.9

17. Secondary Outcome: Change From Baseline in W-BQ22 (Well-being Questionnaire) Index Score at Week 18
Description: The W-BQ22 (well-being) questionnaire was a standardized and generic instrument used for measuring the impact of hypercholesterolemia and treatment on well-being of participants. The general well-being score was calculated as the sum of 22 questions in the W-BQ22 questionnaire (each question scored from 0 to 3 [0 = not at all and 3 = all the time]). Total score for 22 questions range from 0 to 66 [0 = worst condition and 66 = best well-being condition).
Time Frame: From Baseline to Week 18
Population: Analysis was performed on Well-Being analysis set included all randomized and treated participants with complete baseline and complete post-baseline evaluations of the 22-question well-being questionnaire.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 19 | 38
scores on a scale | -1.43 (1.441) | 0.91 (1.04)

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp [a]) (Pre-apheresis) to Week 6
Description: Adjusted means and standard errors at Week 6 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 2 (pre-apheresis) to Week 18 (pre-apheresis) regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percent change | -4 (5.1) | -18.1 (3.7)

19. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) (Pre-apheresis) to Week 6
Description: as for outcome 4
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percent change | 4 (3.4) | 9.3 (2.4)

20. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG) Levels (Pre-apheresis) to Week 6
Description: as for outcome 18
Time Frame: From Baseline to Week 6
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
percent change | 3 (5.6) | -12.9 (4)

21. Secondary Outcome: Percent Change From Baseline in Lp (a) (Pre-apheresis) to Week 18
Description: Adjusted means and standard errors at Week 18 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 2 (pre-apheresis) to Week 18 (pre-apheresis) regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | -1.2 (8) | -6.1 (5.9)

22. Secondary Outcome: Percent Change From Baseline in HDL-C (Pre-apheresis) to Week 18
Description: as for outcome 10
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 2.4 (5) | 10.9 (3.6)

23. Secondary Outcome: Percent Change From Baseline in TG Levels (Pre-apheresis) to Week 18
Description: as for outcome 21
Time Frame: From Baseline to Week 18
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 mg Q2W (Double Blind Period)
Number analyzed (Participants) | 21 | 41
Percent change | 4.1 (7.9) | -2.4 (5.8)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final study end visit (maximum duration: 46 weeks) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs developed/worsened during 'on treatment period'(double blind treatment-emergent period: time from first dose of study drug to last double-blind dose+70 days, prior to first open-label dose of study drug; open-label treatment emergent period: time from first open-label dose of study drug to last dose+70 days).
Groups:
- Placebo Q2W (Double Blind Period): Placebo (for alirocumab) subcutaneous (SC) injection Q2W up to Week 16 (mean exposure of 17 weeks).
- Alirocumab 150 Q2W (Double Blind Period): Alirocumab 150 mg SC injection Q2W up to Week 16 (mean exposure of 17 weeks).
- Alirocumab 150 Q2W (Open Label Treatment Period): Alirocumab 150 mg SC injection Q2W from Week 18 (mean exposure of 17 weeks).
Arm/Group | Placebo Q2W (Double Blind Period) | Alirocumab 150 Q2W (Double Blind Period) | Alirocumab 150 Q2W (Open Label Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/41 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/21 | 4/41 | 1/29
Other Adverse Events (participants affected / at risk) | 10/21 | 22/41 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (Double Blind Period) (N=21) | Alirocumab 150 Q2W (Double Blind Period) (N=41) | Alirocumab 150 Q2W (Open Label Treatment Period) (N=29)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (Double Blind Period) (N=21) | Alirocumab 150 Q2W (Double Blind Period) (N=41) | Alirocumab 150 Q2W (Open Label Treatment Period) (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (4) | 0 (0)
Fatigue (General disorders) | 2 (2) | 6 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.